CLINICAL TRIAL: NCT01093677
Title: A Single-Blind,Randomized,Placebo-Controlled Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Exploratory Pharmacodynamics of LIM-0705 in Male Subjects With Impaired Glucose Tolerance
Brief Title: Investigation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LIM-0705 in Male Subjects With Impaired Glucose Tolerance
Acronym: LIM
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no subjects enrolled
Sponsor: Limerick BioPharma (Industry)
Responsible Party: Wendye Rae Robbins, MD, Limerick BioPharma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIM-0705-CL-003
Record Dates: First submitted 2010-03-15; First posted 2010-03-26 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 750 mg of LIM-0705 BID for 14 days. Up to 20 subjects.
  Interventions: Drug: LIM-0705
- B (Placebo Comparator): Placebo BID for 14 days. Up to 10 subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIM-0705 — Oral solution 750 mg LIM 0705 BID for 14 days.
  Arms: A
Drug: Placebo — Oral solution placebo BID for 14 days.
  Arms: B

SUMMARY:
LIM-0705 will gain results on the effects of LIM-0705 on Male Subjects with Impaired Glucose Tolerance

ELIGIBILITY:
Inclusion Criteria:

1. Males, age 18-70 years old
2. Measured waist circumference to hip circumference ratio >0.90
3. Body mass index (BMI) of 27 - 40 kg/m2
4. Screening and Day -1 capillary glucose measurement between 110-160 mg/dL (6.1-8.9 mmol/L) after a 12 hour fast
5. Screening and Day -1 OGTT with a 2 hour post-glucose measurement ≥140 mg/dL (7.8 mmol/L) after a 12 hour fast
6. Screening HbA1c > 6 and ≤ 7.5%
7. Subjects must be in reasonably good health as determined by pre-study medical history, physical examination, 12-lead ECG, and the following laboratory measures:

   * Electrolytes, ALP, LDH, creatinine, and urea must be within normal range without medication
   * Urinalysis within normal limits
8. Willing to remain in confinement at the clinical study unit for up to 18 days/17 nights and to return to the unit as specified for additional assessments
9. Willing to consume only the food that is provided by the clinical study unit
10. Non-smokers or "social smokers" (defined as fewer than 5 cigarettes per week) willing to abstain from smoking for the duration of study
11. Willing to abstain from alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages
12. Able to read, understand and follow the study instructions
13. Agree to use of two effective methods of contraception

Exclusion Criteria:

1. Allergy to onions or red wine
2. Strict vegetarians (i.e., subjects who do not eat meat, fish, fowl, or dairy)
3. Use of any non-study medication(s) during the study period other than those approved by the Investigator for treatment of an adverse event (AE)
4. Use of chemotherapy agents or history of cancer, other than non-metastatic non-melanoma skin cancer that has been completely excised, within five (5) years prior to the Screening visit
5. Use of any dietary aids or foods known to modulate drug metabolizing enzymes (e.g., St. John's Wort, grapefruit juice) within 4 days of randomization
6. History of bacterial or viral infection requiring treatment with antibiotics or antivirals within 30 days of randomization
7. Difficulty in swallowing oral medications
8. History of seizure disorder
9. Moderate to severe gastro-esophageal reflux disease
10. History of arrhythmia
11. Cognitive or psychiatric disorders, or any other condition that could interfere with compliance with study procedures and/or confinement in a clinical study unit
12. Baseline liver enzymes greater than the upper limit of normal
13. Baseline creatine phosphokinase (CPK) greater than 2.5x the upper limit of normal
14. History of drug or alcohol abuse
15. Use of any other investigational drug within 30 days of randomization or investigational biologic within 180 days of randomization
16. Use of over-the-counter (OTC) medications or nutraceuticals, excluding routine vitamins, within 14 days of randomization or 5 half-lives of the drug, whichever is longer
17. Use of prescription pharmaceuticals within 30 days of randomization
18. Donation and/or receipt of any blood or blood products within 90 days of randomization
19. Current gastrointestinal (GI), renal, hepatic, or coagulant disorder within 12 months of randomization
20. History of peptic or duodenal ulcer or GI bleed
21. Subjects with Gilbert's Syndrome
22. Subjects with positive drug or alcohol screen
23. Subject positive for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of LIM-0705 on glucose metabolism, lipid metabolism and renal function in subjects with impaired glucose tolerance | approx. 1 month
  * Assessment of glucose metabolism will be based on monitoring of overnight-fasting glucose levels and on performance of an Oral Glucose Tolerance Test (OGTT)
  * Assessment of lipid metabolism will be based on 12 hour-fasting lipid profiles (including LDL, HDL, total cholesterol, free fatty acids, and triglycerides)
  * Assessment of renal function will be performed by monitoring serum BUN and creatinine levels

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events and pharmacokinetics of LIM-0705 and its major metabolite | approx. 1 month
  * To evaluate the incidence of treatment emergent adverse events; as well as changes in physical examination findings, vital signs, ECGs, and clinical laboratory tests (serum chemistry, hematology urinalysis, and coagulation)
  * To characterize the pharmacokinetics of LIM-0705 and its major metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Albert Frauman, MD, Study Director — Nucleus Network